CLINICAL TRIAL: NCT02383888
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 425809 in Healthy Japanese and Chinese Male Subjects (Randomized, Double-blind, Placebo-controlled Design Within Dose Groups)
Brief Title: Single Rising Dose Trial of BI 425809 for Healthy Japanese and Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1346.4
Record Dates: First submitted 2015-03-06; First posted 2015-03-10 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

ARMS (4):
- Matching placebo for each dose groups (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 425809 Active dose group 1 (Experimental)
  Interventions: Drug: BI 425809
- BI 425809 Active dose group 2 (Experimental)
  Interventions: Drug: BI 425809
- Bi 425809 Active dose group 3 (Experimental)
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: BI 425809
  Other Names: Iclepertin
  Arms: BI 425809 Active dose group 2
Drug: BI 425809
  Other Names: Iclepertin
  Arms: Bi 425809 Active dose group 3
Drug: Placebo
  Arms: Matching placebo for each dose groups
Drug: BI 425809
  Other Names: Iclepertin
  Arms: BI 425809 Active dose group 1

SUMMARY:
To investigate the safety, tolerability and pharmacokinetics of BI 425809 tablets in healthy Chinese and Japanese male subjects following the administration of single rising oral doses and further to explore the pharmacokinetics (PK) including dose proportionality of BI 425809 after single dosing of product.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age 20 to 45 years (incl.)
* BMI 18.5 to 25 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Chinese ethnicity, Japanese ethnicity according to the following criteria:
* Chinese: ethnic Chinese, born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
* Japanese: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator
* Repeated measurement of systolic blood pressure <90 or >140 mmHg, or diastolic blood pressure <50 or >90 mmHg, or PR <50 or >90
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication
* Diseases of the central nervous system (including by not limited to any kind of seizures or stroke), other neurological disorders or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half- lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* At screening, a marked baseline prolongation of QT/QTcF interval (such as repeated demonstration of a QTcF interval greater than 450 ms or any other relevant ECG finding
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two month after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)
* Evidence or history of macular degeneration or any abnormal finding in color discrimination test, and any other clinically significant ophthalmic disorders based on the investigator's discretion

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the number of subjects with drug-related Adverse Events | up to 18 days post dosing

SECONDARY OUTCOMES:
maximum measured concentration of the analyte in plasma | up to 9 days post doing
area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | up to 9 days post doing
area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable plasma concentration | up to 9 days post doing
time from dosing to the maximum concentration of the analyte in plasma | up to 9 days post doing
terminal half-life of the analyte in plasma | up to 9 days post doing

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1346.4.82001 Boehringer Ingelheim Investigational Site, Busan, South Korea

REFERENCES:
- [Derived] Tsuda Y, Ugai H, Wunderlich G, Shin JG. Pharmacokinetics of Single Doses of BI 425809 in Healthy Chinese and Japanese Subjects: A Randomized Study. Clin Ther. 2019 May;41(5):961-971. doi: 10.1016/j.clinthera.2019.03.014. Epub 2019 Apr 17. PMID 31005336